CLINICAL TRIAL: NCT03511261
Title: Innovative Formulations of Curcumin & Its Comparative Efficacy in Management of Oral Submucous Fibrosis.
Brief Title: Efficacy of Curcumin in Oral Submucous Fibrosis
Acronym: ECOSMF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: H.K.E.S's S.Nijalingappa Institute of Dental Science and Research (Other)
Responsible Party: Principal Investigator, Syeda Arshiya Ara, Professor & Research scholar, H.K.E.S's S.Nijalingappa Institute of Dental Science and Research
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HKESSNDCG/OMR/2014/CT1
Record Dates: First submitted 2017-01-27; First posted 2018-04-27 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Oral Submucous Fibrosis
Keywords: Oral submucous fibrosis; curcumin; potentially malignant disease
MeSH Terms: conditions — Oral Submucous Fibrosis | interventions — Diarylheptanoids; Curcumin

STUDY DESIGN:
Intervention Model Description: four groups, each group with different formulations.
Who Masked: Participant
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- 10%Curcumin mucoadhesive gel (Active Comparator): Drug: Curcumin arm Curcumin10% mucoadhesive gel
  Group 1 patients:
  Drug : 10% curcumin mucoadhesive gel usage : Topical application Frequency : Twice daily Duration : 6 months
  Interventions: Drug: 10% Curcumin mucoadhesive gel
- Curcumin capsules 500mg (Active Comparator): Group 2 patients:
  Drug : curcumin 500 mg capsules usage : oral intake Frequency : Twice daily Duration : 6 months
  Interventions: Drug: Curcumin capsules 500mg
- 5% Curcumin gel+Curcumin capsules 250mg (Active Comparator): Group 3 patients:
  Drug: 5% Curcumin mucoadhesive gel & Curcumin capsules 250mg usage : Topical application and oral intake Frequency : Twice daily Duration : 6 months
  Interventions: Drug: 5% curcumin mucoadhesive gel + Curcumin capsules 250 mg
- Placebo capsules (Placebo Comparator): Group 4 patients Drug: Placebo capsules usage : oral intake Frequency : Twice daily Duration : 6 months
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: 10% Curcumin mucoadhesive gel — Group 1 10%of mucoadhesive gel for topical application two times per day.
  Other Names: curcuminoid
  Arms: 10%Curcumin mucoadhesive gel
Drug: Curcumin capsules 500mg — Group 2 curcumin 500 mg capsules for oral intake two times per day
  Other Names: curcuminoid
  Arms: Curcumin capsules 500mg
Drug: 5% curcumin mucoadhesive gel + Curcumin capsules 250 mg — Group 3 5% curcumin mucoadhesive gel topical application two times per day + curcumin 250 mg capsules for oral intake two times per day
  Other Names: curcuminoid
  Arms: 5% Curcumin gel+Curcumin capsules 250mg
Drug: Placebo capsule — Group 4 placebo capsules for oral intake two times per day
  Other Names: non curcuminoid
  Arms: Placebo capsules

SUMMARY:
The purpose of the study is to determine whether the formulations of curcumin will effect the clinical signs and symptoms and histopathological features in patients with clinical stage 2 oral submucous fibrosis (OSMF).

DETAILED DESCRIPTION:
200 clinical stage 2 OSMF patients selected randomly by simple random technique with clinically & histopathologically confirmed diagnosis are divided into 4 groups with 50 patients each.

In Group 1 patients are given 10% of curcumin mucoadhesive gel and are instructed to use it topically twice daily making it a daily dose of 1gm.

In Group 2 patients are given 500mg of curcumin capsules and are instructed to take 2 capsules twice daily making a daily dose of 1gm.

In Group 3 patients will be given 5% of curcumin mucoadhesive gel and will be instructed to use it topically twice daily & 250mg of curcumin capsules to be taken twice daily making it a daily dose of 1gm.

Group 4 is considered as control group and provided with formulations without the active drug.

The mean scores of 4 groups will be statistically tested using Anova technique.

The differences in clinical parameters at 15 days, 1 month, 3 months & clinical & histopathological paramerters at 6 months will be compared between groups 1, 2, 3 & 4 by using students 't' test & correlation is also used for knowing the association of variables.

For all tests, a 'p' value of 0.05 or less will be utilized for statistical significance.

Other non parametric tests can also be applied where ever necessary for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* 200 clinical stage 2 OSMF patients

Exclusion Criteria:

* Clinical stage 1 & 3 OSMF patients, oromucosal disorders with clinical features same as OSMF, patients who are under treatment, clinically diagnosed cases not ready for incisional biopsy, patients suffering from medically compromised conditions.

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Burning sensation and pain | 6 months for each patient
  Visual Analogue Scale

SECONDARY OUTCOMES:
Interincisal distance, tongue protrusion and cheek flexibility | 6 months for each patient
  All these will be measured in mm at designated time intervals using digital vernier calliper.

CONTACTS AND LOCATIONS:
Overall Officials: Syeda Arshiya Ara, MDS, Principal Investigator — HKE'S S.N Institute of dental sciences & research center
Locations (1):
- HKE'S S.N Institute of dental sciences & research center, Kalaburagi, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hazarey VK, Sakrikar AR, Ganvir SM. Efficacy of curcumin in the treatment for oral submucous fibrosis - A randomized clinical trial. J Oral Maxillofac Pathol. 2015 May-Aug;19(2):145-52. doi: 10.4103/0973-029X.164524. PMID 26604488